CLINICAL TRIAL: NCT00604227
Title: Interstitial Pulmonary Edema After Rapid Ascent to High Altitude (Margherita Hut, 4559 m)
Brief Title: Pulmonary Function at High-Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M2005
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2007-11

CONDITIONS: Pulmonary Edema
Keywords: high altitude pulmonary edema; pulmonary interstitial fluid; pulmonary function testing; hypoxia; pulmonary endothelial function; high altitude exposure without prior acclimatization
MeSH Terms: conditions — Pulmonary Edema; Altitude Sickness; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): high altitude exposure
  Interventions: Other: Hypoxic Exposure

INTERVENTIONS:
Other: Hypoxic Exposure — ascent to 4559 m within 24 h without prior acclimatization

SUMMARY:
Based on the findings of decreased vital capacity, decreased FEV1 and increased closing volume after ascent to high altitude, some investigators suggest the presence of a subclinical high altitude pulmonary edema (HAPE). Since these parameters are only indirect measures of pulmonary interstitial fluid accumulation, the aim of this study is to examine the effects of broncho-constriction on the increase of closing volume by extensive lung function testing in healthy mountaineers at low altitude and on the Margherita Hut (4559 m). As has been done in earlier studies, conventional thorax radiographs are used for verification of HAPE. In this study, the determination of the thoracic fluid quantity will be completed by measurements of thoracic impedance. In addition markers of pulmonary endothelial function will be assessed to get further insight into the regulation of pulmonary vascular tone at altitude and in particular into the pathophysiology of HAPE.

ELIGIBILITY:
Inclusion Criteria:

* Mountaineering ability required for reaching the Margherita hut (4559 m)

Exclusion Criteria:

* Borne above 1500 m
* Subjects with internal medical diseases like all cardiac diseases, all pulmonary diseases, Diabetes mellitus, infectious diseases, thyroid diseases, malignant diseases, hepatic or renal diseases,
* (Known) hypersensitivity to salbutamol or to another component of sultanol® or lidocaine, or to another component of xylocain® pump spray
* Intake of drugs, especially nifedipine, acetazolamide and glucocorticoids or of drugs interacting with sultanol® or xylocain® pump spray
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2005-07; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
development of HAPE | during the 48 h stay at altitude

SECONDARY OUTCOMES:
change of lung function parameters from low to high altitude | during the 48 h stay at altitude
markers of pulmonary endothelial function | during the 48 h stay at altitude
quantification of pulmonary interstitial fluid | during the 48 h stay at altitude

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Dehnert, MD, Principal Investigator — University Hospital Heidelberg; Marc M Berger, MD, Principal Investigator — University Hospital Heidelberg; Peter Bärtsch, MD, PhD, Study Director — University Hospital Heidelberg
Locations (1):
- Sports Medicine, University Hospital, Heidelberg, Germany